CLINICAL TRIAL: NCT00066443
Title: A Phase I/II Study Of Increasing Doses Of Epirubicin And Docetaxel Plus Pegfilgrastim For Locally Advanced Or Inflammatory Breast Cancer
Brief Title: Epirubicin, Docetaxel, and Pegfilgrastim in Treating Women With Locally Advanced or Inflammatory Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA22; CAN-NCIC-MA22; CDR0000316237 (Other: PDQ)
Record Dates: First submitted 2003-08-06; First posted 2003-08-07 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer
Keywords: stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; inflammatory breast cancer
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms | interventions — pegfilgrastim; Docetaxel; Epirubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pegfilgrastim, docetaxel and epirubicin (Experimental)
  Interventions: Biological: pegfilgrastim; Drug: docetaxel; Drug: epirubicin hydrochloride

INTERVENTIONS:
Biological: pegfilgrastim — Dose escalation schedule A&B = 6mg fixed dose once per cycle on day 2
Drug: docetaxel — Dose Escalation schedule A = 75-85 mg/m2 Dose Escalation schedule B = 50-75 mg/m2
Drug: epirubicin hydrochloride — Dose escalation schedule A = 75-120 mg/m2 IV Dose escalation schedule B = 50-90 mg/m2 IV

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as epirubicin and docetaxel use different ways to stop tumor cells from dividing so they stop growing or die. Colony-stimulating factors such as pegfilgrastim may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of chemotherapy.

PURPOSE: Phase I/II trial to study the effectiveness of combining epirubicin and docetaxel with pegfilgrastim in treating women who have locally advanced or inflammatory breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and recommended phase II dose of docetaxel and epirubicin when given with pegfilgrastim in women with locally advanced or inflammatory breast cancer. (Phase I, group 1 closed to accrual as of 9/13/04 and Phase II, group 1 closed to accrual as of 5/10/06)
* Determine the toxicity of this regimen in these patients.
* Determine the clinical and pathological response rate and duration of response in patients treated with this regimen.
* Determine drug sensitivity and resistance in patients treated with this regimen.
* Determine prognostic and predictive markers in patients treated with this regimen.

OUTLINE: This is a nonrandomized, multicenter, dose-escalation study of docetaxel and epirubicin.

* Phase I:

Group 1 (21-day regimen) (closed to accrual as of 09/13/04): Patients receive epirubicin IV over 15 minutes and docetaxel IV over 60 minutes on day 1 and pegfilgrastim subcutaneously on day 2. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients with objective response after 6 courses may receive additional therapy at the discretion of the physician.

Group 2 (14-day regimen): Patients receive epirubicin IV over 15 minutes and docetaxel IV over 60 minutes on day 1 and pegfilgrastim subcutaneously on day 2. Treatment repeats every 14 days for up to 8 courses in the absence of disease progression or unacceptable toxicity. Patients with objective response after 8 courses may receive additional therapy at the discretion of the physician.

Cohorts of 3-6 patients receive escalating doses of epirubicin and docetaxel until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

* Phase II:

Group 1 (21-day regimen) (closed to accrual as of 5/10/06): Patients receive treatment as in phase I with epirubicin and docetaxel at the recommended Phase II dose.

Group 2 (14-day regimen): Patients receive treatment as in phase I with epirubicin and docetaxel at the recommended Phase II dose.

Patients are followed at 1 month, every 3 months for 1 year, every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 90 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive adenocarcinoma of the breast, meeting any of the following criteria:

  * T4, NX, M0
  * Any T, N2-N3, M0
  * Inflammatory breast cancer (redness over at least one-third of the breast), M0
* No evidence of metastatic disease by chest x-ray, abdominal ultrasound or CT scan and bone scan
* Diagnosed within the past 8 weeks
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 16 and over

Sex

* Female

Menopausal status

* Not specified

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute granulocyte count at least 2,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic

* Bilirubin less than upper limit of normal (ULN)
* Must meet criteria for 1 of the following:

  * ALT and AST no greater than 1.5 times ULN AND alkaline phosphatase no greater than 2.5 times ULN
  * ALT and AST normal AND alkaline phosphatase no greater than 5 times ULN

Renal

* Creatinine no greater than 1.5 times ULN

Cardiovascular

* Resting LVEF normal by MUGA or echocardiogram
* No congestive heart failure
* No angina pectoris
* No myocardial infarction within the past year
* No uncontrolled hypertension
* No uncontrolled arrhythmias

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective non-hormonal contraception
* No other malignancy within the past 5 years except adequately treated nonmelanoma skin cancer or curatively treated carcinoma in situ of the cervix
* No symptomatic peripheral neuropathy grade 2 or greater
* No active infection
* No history of significant neurological or psychiatric disorders, including dementia or seizures
* No peptic ulcer
* No unstable diabetes mellitus
* No contraindication to dexamethasone
* No known sensitivity to E. coli-derived or polyethylene glycol products
* Willing to undergo core biopsies once prior to registration and core biopsies at 2 other timepoints while on study
* Geographically accessible for treatment and follow-up

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior immunotherapy for breast cancer

Chemotherapy

* No prior chemotherapy for breast cancer

Endocrine therapy

* No prior hormonal therapy for breast cancer
* No concurrent corticosteroids except for premedication or hypersensitivity reaction
* No concurrent oral contraception

Radiotherapy

* No prior radiotherapy for breast cancer

Surgery

* No prior surgery for breast cancer other than biopsy

Other

* No prior systemic therapy for breast cancer
* No other concurrent investigational drugs or anticancer treatment
* No concurrent preventative IV antibiotics

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2003-11-03 (Actual); Primary Completion 2010-01-06 (Actual); Study Completion 2014-01-16 (Actual)

PRIMARY OUTCOMES:
Toxic effects | 7 years
  Findings were presented at ASCO 2010
Response (phase II) | 12 years
  Response was presented at ASCO 2010. Duration of response will be analyzed in 2015

CONTACTS AND LOCATIONS:
Overall Officials: Maureen E. Trudeau, BSc, MA, MD, FRCPC, Study Chair — Toronto Sunnybrook Regional Cancer Centre
Locations (5):
- Canada (5):
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Atlantic Health Sciences Corporation, Saint John, New Brunswick
  - Odette Cancer Centre, Toronto, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CHA-Hopital Du St-Sacrement, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Yes
URL: https://www.ctg.queensu.ca/docs/public/policies/DataSharingandAccessPolicy.pdf

REFERENCES:
- [Result] Parissenti AM, Chapman JA, Kahn HJ, Guo B, Han L, O'Brien P, Clemons MP, Jong R, Dent R, Fitzgerald B, Pritchard KI, Shepherd LE, Trudeau ME. Association of low tumor RNA integrity with response to chemotherapy in breast cancer patients. Breast Cancer Res Treat. 2010 Jan;119(2):347-56. doi: 10.1007/s10549-009-0531-x. PMID 19771508
- [Result] Trudeau ME, Chapman JA, Guo B, Clemons MJ, Dent RA, Jong RA, Kahn HJ, Pritchard KI, Han L, O'Brien P, Shepherd LE, Parissenti AM. A phase I/II trial of epirubicin and docetaxel in locally advanced breast cancer (LABC) on 2-weekly or 3-weekly schedules: NCIC CTG MA.22. Springerplus. 2015 Oct 21;4:631. doi: 10.1186/s40064-015-1392-x. eCollection 2015. PMID 26543765
- [Derived] Parissenti AM, Guo B, Pritzker LB, Pritzker KP, Wang X, Zhu M, Shepherd LE, Trudeau ME. Tumor RNA disruption predicts survival benefit from breast cancer chemotherapy. Breast Cancer Res Treat. 2015 Aug;153(1):135-44. doi: 10.1007/s10549-015-3498-9. Epub 2015 Jul 25. PMID 26208483
- [Derived] Pritzker K, Pritzker L, Generali D, Bottini A, Cappelletti MR, Guo B, Parissenti A, Trudeau M. RNA Disruption and Drug Response in Breast Cancer Primary Systemic Therapy. J Natl Cancer Inst Monogr. 2015 May;2015(51):76-80. doi: 10.1093/jncimonographs/lgv015. PMID 26063893